CLINICAL TRIAL: NCT02332018
Title: Two-dimensional And Three-dimensional Measurements Of Torsion And Length Of Lower Limbs And Spine Based On Biplanar Radiographs: Microdose Imaging Protocol Compared To Standard Dose Imaging Protocol
Brief Title: Measurements Of Lower Limbs And Spine Based On Biplanar Radiographs: Microdose Compared To Standard Dose Protocol
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr.: 2014-0405
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Underdevelopment; Congenital Malformation, Lower Limb; Scoliosis
MeSH Terms: conditions — Congenital Abnormalities; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Limb Torsion: adult patients, lower limb assessment retrospectively limb length and limb axis, torsion biplanar x-ray images
  Interventions: Radiation: Biplanar x-ray images
- Limb Length and Axis: adult patients, lower limb assessment prospectively limb length and limb axis biplanar x-ray images
  Interventions: Radiation: Biplanar x-ray images
- Spine: adult patients, spine assessment prospectively Cobb angles, plumbline biplanar x-ray images
  Interventions: Radiation: Biplanar x-ray images

INTERVENTIONS:
Radiation: Biplanar x-ray images — biplanar x-ray images with microdose and low-dose protocol

SUMMARY:
Evaluation of accuracy and reliability of 2D and 3D measurements of the spine and lower limbs in adults based on biplanar radiographs with MicroDose protocol compared to a standard dose protocol

DETAILED DESCRIPTION:
Evaluation of accuracy and reliability of 2D and 3D measurements of the spine and lower limbs in adults based on biplanar radiographs with MicroDose protocol compared to a standard dose protocol

Part 1: retrospective evaluation of 50 patients: lower limb images with MicroDose protocol and lower limb images with standard dose protocol Part 2: prospective evaluation of 100 patients: lower limb images with MicroDose protocol and lower limb images with standard dose protocol Part 3: prospective evaluation of 150 patients: spine images with MicroDose protocol and spine limb images with standard dose protocol

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: All patients referred for biplanar radiographs of spine and lower limb (from 18 to 99 years of age)

Exclusion Criteria:

* Exclusion criteria: no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients referred for assessment of spine or lower limb with biplanar x-ray-scanner
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

PRIMARY OUTCOMES:
2D- and 3D- measurements (torsion angles, scoliotic and kyphotic angles, length etc.) on biplanar radiographs with and without "MicroDose"-protocol and comparison of image quality parameters | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rosskopf, Principal Investigator — Balgrist University Hospital
Locations (1):
- Radiology Department, Balgrist University Clinic, Zurich, Canton of Zurich, Switzerland